CLINICAL TRIAL: NCT04376944
Title: Evaluating Effectiveness of Barrier Measures to Limit Nosocomial Transmission: Covid-19 Prevalence Survey Among Caregivers With Various Exposures
Brief Title: Barrier Measures to Limit Covid-19.Nosocomial Transmission: a Cross-sectional Evaluation
Acronym: EMBELLIE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0261
Record Dates: First submitted 2020-05-04; First posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Caregivers; COVID-19
Keywords: barrier measures
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — NC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed group: Caregivers and agents working directly in COVID units compared to those living.
  Interventions: Other: Survey
- Control group: caregivers anf agents working in services excluding the management of patients screened positive for Covid-19 infection
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — questionnaire on their symptoms and their exposures

SUMMARY:
Use lay language. The Covid-19 pandemic hit France in March 2020 and stage 3 of the epidemic justified the introduction of national and unprecedented containment measures from March 17, 2020. The Montpellier CHU experienced peak hospitalizations of Covid-19 infections in late March. The estimate of the proportion of infected people in Occitania, South of France, for the 11th of May 2020 is 3.1% (95% CI: 1.9-5.9) for the Occitania region, to which Montpellier belongs.

In the context of the Covid-19 epidemic, notably due to the absence of pharmacological or vaccine prophylaxis, barrier measures were of crucial importance, especially for exposed caregivers. These measures include an adaptation of individual behavior, the creation of a so-called "Covid" hospital, the wearing of specific equipment in all departments, the use in the rooms of Covid-19 patients of a gown, an apron, gloves, and a FFP2 type mask in the event of contact and sampling, protocolized and standardized bio-cleaning measures, a reorganization of the premises and the definition of specific circuits.

In view of the second wave of the epidemic, estimating the effectiveness of the barrier measures is of major importance. The investigators therefore propose an evaluation of the effectiveness of these measures, by comparing the serological prevalence of infection among caregivers working directly in COVID units compared to caregivers working in services excluding the management of Covid-19 patients.

Systematic evaluation in COVID-19 units of Sarc-Co-V2 infection will also be assessed, with naso-pharyngeal swabs.

ELIGIBILITY:
Inclusion criteria:

* exposed group: exposed caregivers and agents who worked in COVID units (medicine, resuscitation, screening) until their date of collection. An exposed agent or caregiver is defined by the entrance of rooms with a COVID-19 infection during their professional activity.
* low or unexposed group: caregivers or agents who have worked in non-COVID units in a non-COVID hospital

Exclusion criteria:

- refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: carers of the UH Montpellier
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of caregivers and agents with a positive serodiagnosis | 1 day
  Proportion of caregivers and agents with a positive serodiagnosis in COVID units versus non-COVID units

SECONDARY OUTCOMES:
Proportion of caregivers and agents with a positive RT-PCR | 1 day
  Proportion of caregivers and agents with a positive RT-PCR in COVID units versus non-COVID units

CONTACTS AND LOCATIONS:
Overall Officials: Marie Bistoquet, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC